CLINICAL TRIAL: NCT03930706
Title: Clinical Pregnancy Rate for Frozen Embryo Transfer With Hormonal Replacement Therapy (HRT): a Pilot Study Comparing 1 Versus 2 Weeks of Treatment
Brief Title: SHorter Treatment of Replacement Therapy for Frozen Embryo Transfer (FET)
Acronym: ShoRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Blockeel Christophe, Professor Doctor, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRT1vs2week.2018
Record Dates: First submitted 2019-04-16; First posted 2019-04-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Group A will include all the patient that will start with progesterone ((P), Utrogestan®) supplementation after 7 days of E2 (Progynova®) intake and that will perform the FET (after 13 days of E2 and 6 days of P).
  Interventions: Other: Longer administration of estradiol (Progynova®)
- Group B (Active Comparator): Group B will include the patients that will perform 14 days of E2 intake (Progynova®, 6 mg per day (2 mg every 8 hours) those patients will be asked to perform a supplementary blood test and ultrasound on day 14 of E2 intake, afterwards, they will start with P supplementation (Utrogestan®, 800 mg per day, 400 mg every 12 hours) from day 15 of E2 for 6 days and they will get their FET day 20 of the cycle (after 14 days of E2 and 6 days of P)
  Interventions: Other: Longer administration of estradiol (Progynova®)

INTERVENTIONS:
Other: Longer administration of estradiol (Progynova®) — All women included will take exogenous hormone with daily administration of Estradiol Valerate (Progynova®), the standard dose used will be 6 mg/day (Cobo et al., n.d.). On day 7 of endometrial preparation patients will be examined with vaginal ultrasound and blood test, to evaluate the endometrial thickness and the hormones levels. In both arms the FET will take place after 6 days of Progesterone supplementation (600 mg per day, vaginal administration of Utrogestan®) According to embryo quality after warming, embryo transfer to the uterine cavity will be performed on day 5 of development under ultrasound guidance whenever possible. Following embryo transfer, luteal support will be continued with vaginally administered P (Utrogestan®). All patients 12 days after the FET will undergo the pregnancy test (blood test to evaluate hCG).
  Other Names: comparing 7 vs 14 days of administration of estradiol (Progynova®) for artificially prepared endometrium in frozen embryo transfer

SUMMARY:
This is a Single-centre pilot study, randomized, controlled open-label trial with the aim to assess the clinical pregnancy rate and the early pregnancy loss rate between two different schemas for frozen embryo transfer cycles stimulated with HRT. Furthermore, the investigators would like to evaluate the predictivity of pregnancy and early miscarriage by looking at the endocrinological profile (estradiol and progesterone levels) within the endometrial preparation and the day of embryo transfer (ET).

DETAILED DESCRIPTION:
Women planned for a FET-HRT will be asked to do a blood test day 1 of their cycle in order to evaluate the endocrine profile; those with basal hormonal values will receive 6 mg oral estradiol daily beginning from day 1 of their cycle. On day 7 of the treatment a blood test for the serum hormone evaluation and an ultrasound will be planned in order to evaluate the endometrium thickness; those who will meet the criteria (endometrium thickness ≥7mm) will be randomized. In the 7 days estradiol (E2) arm (A) the study coordinator will plan the FET after 6 days of progesterone supplementation (13 days of E2 intake). In the 14 days E2 arm (B) the team will plan on day 14 of treatment with E2 the serum hormone evaluation and an ultrasound in order to evaluate the endometrium thickness, consequently the FET will be planned after 6 days of progesterone supplementation (after 14 days of E2 intake). Furthermore, all the patients included in the study will undergo a blood test on the day of the transfer for the evaluation of the hormones level. For the assessment of the pregnancy a first blood test will take place 12 days after the ET and a blood test with an ultrasound will take place at 7 weeks for the evaluation of the clinical pregnancy.

ELIGIBILITY:
* Women aged ≥18 and < 40 years
* Unexplained infertility
* Normal uterine cavity
* IVF/ICSI
* IVF cycle with GnRH agonist or antagonist
* Single day 5 blastocyst transfer
* Top quality embryo (at least Bl 3BA) at the moment of ET
* Signed informed consent
* Participants can be included only once in the trial
* Informed consent documents signed prior to screening evalua-tions.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate | 2 years
  The number of clinical pregnancies expressed per 100 initiated cycles, aspiration cycles or embryo transfer cycles. When clinical pregnancy rates are recorded, the denominator (initiated, aspirated or embryo transfer cycles) must be specified.
Live Birth Rate | 4 years
  The number of deliveries that resulted in at least one live birth, expressed per 100 cycle attempts. In the case of assisted reproductive technologies (ART) interventions, they can be initiated cycles, insemination, aspiration cycles or embryo transfer cycles. When delivery rates are given, the denominator (initiated, inseminated, aspirated or embryo transfer cycles) must be specified.
Miscarriage rate | 2 years
  The spontaneous loss of an intra-uterine pregnancy prior to 22 completed weeks of gestational age, over the number of transferred embryos.

SECONDARY OUTCOMES:
positive hCG tests | 2 years
  the number of participants with positive hCG measured on a blood sample 12 days after ET
biochemical pregnancy | 2 years
  the number of patients with positive hCG but no embryo development assessed
early pregnancy loss | 2 years
  the number of participants who had a pregnancy loss before 8 weeks of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Blockeel, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

REFERENCES:
- [Derived] Racca A, Santos-Ribeiro S, Drakopoulos P, De Coppel J, Van Landuyt L, Tournaye H, Blockeel C. Clinical pregnancy rate for frozen embryo transfer with HRT: a randomized controlled pilot study comparing 1 week versus 2 weeks of oestradiol priming. Reprod Biol Endocrinol. 2023 Jul 7;21(1):62. doi: 10.1186/s12958-023-01111-8. PMID 37420186